CLINICAL TRIAL: NCT01226446
Title: Multicenter Open and Prospective Trial Assessing the Efficacy of Vitamin D Supplementation in Addition to Pegylated Interferon Plus Ribavirin in Null-Responders Patients With Chronic Viral Hepatitis C Genotype 1 or 4
Brief Title: Efficacy of Vitamin D on Top of Pegylated Interferon and Ribavirin in Patients With Chronic Viral Hepatitis C Null-Responders
Acronym: ANRS VITAVIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021967-34
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Addition of Vitamin D to Peg-interferon plus Ribavirin (Experimental)
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: vitamin D — Vitamin D on top of the standard treatment

SUMMARY:
Vitamin D deficiency is commonly found in patients with chronic hepatitis C. The investigators hypothesize that the correction of hypovitaminosis D before the initiation of anti-HCV combination therapy and the maintenance of an optimal vitamin D status during antiviral therapy could improve the antiviral efficacy

DETAILED DESCRIPTION:
An open-label, prospective evaluation of the efficacy of vitamin D supplementation starting 1 month before and continuing for the duration of combination therapy with pegylated interferon alpha (2a or 2b) plus ribavirin in patients with chronic viral hepatitis C genotype 1 or 4, nonresponders to a first antiviral therapy.Vitamin D supplementation is started one month before antiviral therapy in order to introduce pegylated interferon plus ribavirin in patients with optimal vitamin D status

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C Genotype 1 or 4
* Hypovitaminosis D defined by a value <30 ng / ml
* Patient non responder to previous antiviral combination therapy of Pegylated Interferon and Ribavirin defined by a decrease in viral load <2 log at week 12 of the first course (Peg/RBV)
* Patient who received at least 80% of the optimal dose of Pegylated Interferon and Ribavirin according to current recommendations
* Patient for which the investigating physician decided to initiate treatment for hepatitis C combination therapy

Exclusion Criteria:

* Decompensated liver disease: Child-Pugh B> 8 or one of the following criteria: bilirubin> 35 micromol/L, TP <50%, ascites, recurrent encephalopathy
* Positive serology for HBV and HIV
* Alcohol consumption exceeding 50 g/day
* Chronic intake of vitamin D
* Thrombocytopenia <50 000/mm ³, neutropenia <750/mm ³, hemoglobin <11 g/dL
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Negativity of HCV RNA below 12UI/mL after 12 weeks of antiviral combination therapy | at week 12

SECONDARY OUTCOMES:
Changes in HCV viral load after correction of vitamin D deficiency (delta log) | at day 0
Changes in HCV viral load (delta log) | at week 4
Changes in HCV viral load (delta log) | at week 12
Negativity of HCV RNA below 12 UI/ml | at week 24
Negativity of HCV RNA below 12 UI/ml | at week 72

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Cacoub, MD, Principal Investigator — Pitié Salpétrière Hospital
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Terrier B, Lapidus N, Pol S, Serfaty L, Ratziu V, Asselah T, Thibault V, Souberbielle JC, Carrat F, Cacoub P. Vitamin D in addition to peg-interferon-alpha/ribavirin in chronic hepatitis C virus infection: ANRS-HC25-VITAVIC study. World J Gastroenterol. 2015 May 14;21(18):5647-53. doi: 10.3748/wjg.v21.i18.5647. PMID 25987791